CLINICAL TRIAL: NCT03681574
Title: Use of Gabapentin as Preanesthetic Medication in Oncologic Children Undergoing in Fast Procedures With Sevofluran
Brief Title: Gabapentin as Preanesthetic Medication to Fast Procedures in Pediatric´s Oncology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Infantil Albert Sabin (Other)
Responsible Party: Principal Investigator, washington aspilicueta pinto filho, Principal Investigator, anesthetist, Hospital Infantil Albert Sabin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOSPITALIAS2
Record Dates: First submitted 2018-09-11; First posted 2018-09-24 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Pain, Postoperative; Agitation States as Acute Reaction to Exceptional Stress; Anesthesia; Vomiting
Keywords: pediatric; gabapentin; agitation; induction
MeSH Terms: conditions — Pain, Postoperative; Vomiting; Psychomotor Agitation | interventions — Spinal Puncture; Myelography; gamma-Aminobutyric Acid; Population Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: A pharmacist will prepare the drugs under codes of numbers 1, 2 or 3. The nursing team and anesthesiologists will not know the drug formula used. Drugs will only be revealed after the statistical assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Group (Experimental): The placebo group will receive placebo concentrate orally (0.3 mL/kg) only once, 1 to 2 hours before the oncologic procedure. All patients will undergo the same anesthetic protocol. Afterward, the patients will be submitted to oncologic procedures: Myelogram or Lumbar Puncture.
  Interventions: Drug: Placebo Group
- GABA 15mg/kg Group (Experimental): The GABA 15mg/kg group will receive gabapentin syrup orally (15 mg/kg) only once, 1 to 2 hours before the oncologic procedure. All patients will undergo the same anesthetic protocol. Afterward, the patients will be submitted to oncologic procedures: Myelogram or Lumbar Puncture.
  Interventions: Drug: GABA 15mg/kg Group
- GABA 30mg/kg Group (Experimental): The GABA 30mg/kg group will receive gabapentin syrup orally (30 mg/kg) only once, 1 to 2 hours before the oncologic procedure. All patients will undergo the same anesthetic protocol. Afterward, the patients will be submitted to oncologic procedures: Myelogram or Lumbar Puncture.
  Interventions: Drug: GABA 30mg/kg Group

INTERVENTIONS:
Drug: Placebo Group — Patients will be submitted to either myelogram or lumbar puncture procedure. Before that they will receive placebo concentrate.
  Other Names: Lumbar puncture; Myelogram
  Arms: Placebo Group
Drug: GABA 15mg/kg Group — Patients will be submitted to either myelogram or lumbar puncture procedure. Before that they will receive gabapentin at 15mg/kg.
  Other Names: Lumbar puncture; Myelogram
  Arms: GABA 15mg/kg Group
Drug: GABA 30mg/kg Group — Patients will be submitted to either myelogram or lumbar puncture procedure. Before that they will receive gabapentin at 30mg/kg.
  Other Names: Lumbar puncture; Myelogram
  Arms: GABA 30mg/kg Group

SUMMARY:
This study is a clinical trial, prospective, randomized and double-blinded. Placebo, Gabapentin syrup at 15 mg/kg, and Gabapentin syrup at 30 mg/kg were administered to reduce agitation before and after in children submitted procedures (myelogram or lumbar puncture) among 1 and 6 years.

DETAILED DESCRIPTION:
Gabapentin syrup at 15 mg/kg and at 30 mg/kg was administered to reduce the agitation before and after oncologic procedures (myelogram or lumbar puncture) in children among 1 and 6 years. Three groups were compared: the control group received placebo, the other two groups received gabapentin at 15mg/kg or at 30mg/kg. All patients received the same protocols (anesthesia and analgesia). Anesthesia protocol used was induction with sevoflurane 8% plus N2O 50% and oxygen, maintenance with sevoflurane 4%. We provided local analgesia with 5% lidocaine creme before the procedure. If it was required, dipyrone 10mg/kg every 6 hours was given as rescue analgesia. To prevent post-operative vomit, ondasentron 0,1mg/kg was administered when intrathecal chemotherapy. The mYPAS scale was used to evaluate preoperative anxiety at several moments: at basal, at after 1-hour administration, at separation from parents, and at induction. The PAED scale was applied after 30 minutes of procedure to evaluate postoperative agitation. The CHIPPS scale was used to assess postoperative pain. The frequency of vomits was recorded for 8 hours after the procedure finished.

ELIGIBILITY:
Inclusion Criteria:

* Cancer or under investigation for cancer.
* Children between 1 and 6 years.
* Previously submitted to oncologic procedures, e.g. myelogram or puncture lumbar.

Exclusion Criteria:

* Cardiac disease.
* Pulmonary disease.
* Renal disease.
* Neurological disease.
* Any allergies.
* Refusal of parents, caregivers or patients to participate in the study.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
The intensity of anxiety in children by Modified Yale Preoperative Anxiety Scale (mYPAS) before an oncologic procedure under Gabapentin or placebo effects. | 8 hours
  Children, ranging from 1 to 6 years old, will receive drugs (placebo, gabapentin 15mg/kg or 30mg/kg) 1 to 2 hours before the oncologic procedure (myelogram and/ or puncture lumbar). They will be submitted to the same general anesthesia protocol (sevoflurane 8% plus N2O and oxygen) and postoperative analgesia. All patients will be observed for changes in the Modified Yale Preoperative Anxiety Scale (mYPAS) at baseline (right before drug administration), at 1 hour after group administration, at the separation from parents, and at anesthetic induction time. The mYPAS scale is a compilation of 5 subscales: activity (0 to 4 points), vocalizations (0 to 6 points), emotional expressivity (0 to 4 points), state of apparent arousal (0 to 4 points), and use of parent (0 to 4 points). All scores are summed up, divided by 4, and then multiplied by 100. Total scores above 30 points are interpreted as a patient with anxiety, which would represent a worse outcome.

SECONDARY OUTCOMES:
Percentage of sevoflurane consumption in patients over anesthetic induction. | 8 hours
  Patients will be submitted to the same general anesthesia protocol, receiving sevoflurane 8% plus N2O and oxygen prior to the procedure. We will measure the percentage of sevoflurane ended-expired.
Level of emergence delirium and agitation in children at post-operative through Paediatric Anaesthesia Emergence Delirium. | 1 hour
  After the procedure, all patients will be observed for change in the Paediatric Anaesthesia Emergence Delirium (PAED 0 to 20 points) scale. Score changes will be assessed at baseline (right after the procedure), and at 30 minutes the procedure has finished. Each criterion is assessed through the event frequency, e.g. "eye contact" that "never" occurs corresponds to score 4. The range goes from "never" (4 points) up to "always" (0 points) for positive behavior criteria. Those are "make contact with the caregiver", "actions are purposeful", and "aware of surroundings". Negative behavior criteria range from "never" (0 points) up to "always" (4 points). Those are "restlessness" and "inconsolable". All subscores are summed up into a total score. Total scores above 10 points are interpreted as a patient with emergence delirium, which would indicate a worse outcome.
Frequency of post-operative vomits. | 8 hours
  All patients will be evaluated number of vomits occurrence for 8 hours after procedure.
Anesthetic induction time in seconds. | 8 hours
  Patients will be submitted to the same general anesthesia protocol, receiving sevoflurane 8% plus N2O and oxygen prior to the procedure. We will record the time, in seconds, when patients lose their consciousness and corneal reflex.
Levels of postoperative pain in children through Children and Infants Postoperative Pain Scale (CHIPPS). | 1 hour
  After the procedure, all patients will be observed for changes in the Children and Infants Postoperative Pain Scale (CHIPPS) scores. Score changes will be assessed at baseline (right after the procedure), and at 30 minutes the procedure has finished. The score ranges from 0 (Behavior not present) to 2 (Intense behavior), to be assessed in each of the following indicators: "crying", "facial expression", "posture of the trunk", "posture of legs", and "motor restlessness". All subscores are summed up into a total score. Total scores above 6 points are interpreted as a patient with severe pain, which would indicate a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil Albert Sabin, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rusy LM, Hainsworth KR, Nelson TJ, Czarnecki ML, Tassone JC, Thometz JG, Lyon RM, Berens RJ, Weisman SJ. Gabapentin use in pediatric spinal fusion patients: a randomized, double-blind, controlled trial. Anesth Analg. 2010 May 1;110(5):1393-8. doi: 10.1213/ANE.0b013e3181d41dc2. PMID 20418301
- [Result] Mayell A, Srinivasan I, Campbell F, Peliowski A. Analgesic effects of gabapentin after scoliosis surgery in children: a randomized controlled trial. Paediatr Anaesth. 2014 Dec;24(12):1239-44. doi: 10.1111/pan.12524. Epub 2014 Sep 17. PMID 25230144
- Available data/document: Study Protocol: study protocol — https://www.justbeamit.com/k7ciq — study protocol
- Available data/document: Individual Participant Data Set: data set — https://www.justbeamit.com/nwxjr — individual participant data set
- Available data/document: Informed Consent Form: informed consent form — https://www.justbeamit.com/n2c2d — consert form
- Available data/document: Statistical Analysis Plan: statistical plan — https://www.justbeamit.com/43kxq — statistical plan